CLINICAL TRIAL: NCT03156842
Title: A Randomized, Double-blind, Multicenter, Phase III Study to Evaluate the Efficacy and Safety of Combination Treatment of Fimasartan/Amlodipine/Rosuvastatin in Patients With Essential Hypertension and Dyslipidemia Who Fail to Respond Adequately to Fimasartan Monotherapy
Brief Title: Combination of Fimasartan/Amlodipine/Rosuvastatin in Patients With Essential Hypertension and Dyslipidemia
Acronym: FIRST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BR-FARC-CT-301
Record Dates: First submitted 2017-05-14; First posted 2017-05-17 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Essential Hypertension; Dyslipidemia
Keywords: Hypertension; Dyslipidemia; Fimasartan; Rosuvastatin
MeSH Terms: conditions — Essential Hypertension; Dyslipidemias; Hypertension | interventions — fimasartan; Amlodipine; Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fimasartan/Amlodipine, Rosuvastatin (Experimental): Co-administration of a fixed dose combination of Fimasartan/Amlodipine and Rosuvastatin
  Interventions: Drug: Fimasartan/Amlodipine, Rosuvastatin
- Fimasartan/Amlodipine (Active Comparator): a fixed dose combination of Fimasartan/Amlodipine
  Interventions: Drug: Fimasartan/Amlodipine
- Fimasartan, Rosuvastatin (Active Comparator): Co-administration of Fimasartan and Rosuvastatin
  Interventions: Drug: Fimasartan, Rosuvastatin

INTERVENTIONS:
Drug: Fimasartan/Amlodipine, Rosuvastatin — "A fixed dose combination tablet of Fimasartan and Amlodipine" and "Rosuvastatin" will be administrated once daily on treatment period.
  Arms: Fimasartan/Amlodipine, Rosuvastatin
Drug: Fimasartan/Amlodipine — "A fixed dose combination tablet of Fimasartan and Amlodipine" will be administrated once daily on treatment period.
  Arms: Fimasartan/Amlodipine
Drug: Fimasartan, Rosuvastatin — "Fimasartan" and "Rosuvastatin" will be administrated once daily on treatment period.
  Arms: Fimasartan, Rosuvastatin

SUMMARY:
The objective of this clinical study is to evaluate the efficacy and safety by comparing the fimasartan/amlodipine/rosuvastatin treatment group to the fimasartan/amlodipine treatment group and the fimasartan/rosuvastatin treatment group respectively at Week 8 in patients with essential hypertension and dyslipidemia who fail to respond to the fimasartan monotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily provided a written consent to participate in this clinical study
2. Male or female adults aged 19-70 years
3. Patients must have been confirmed essential hypertension and dyslipidemia at Screening visit (V1)
4. Uncontrolled blood pressure (140 mmHg ≤ mean Sitting systolic blood pressure(SiSBP) < 180 mmHg) at the baseline visit (V3) after the fimasartan 60 mg monotherapy
5. Subjects who meet the following criteria of fasting serum lipid levels confirmed at the baseline visit (V3) after undergoing the therapeutic lifestyle change (TLC)
6. Treatment compliance of fimasartan 60 mg ≥70% at the baseline visit (V3)
7. Able to understand this study, be cooperative in the execution of the study, and participate in the study until its completion

Exclusion Criteria:

1. Severe hypertension with mean Sitting systolic blood pressure(SiSBP) ≥180 mmHg or Sitting diastolic blood pressure(SiDBP) ≥110 mmHg at the screening visit (V1) and the baseline visit (V2, or orthostatic hypotension accompanied by symptoms
2. Differences between arms greater than 20 mmHg for Sitting systolic blood pressure(SiSBP) and 10 mmHg for Sitting diastolic blood pressure(SiDBP) are present on 3 consecutive readings at the screening visit (V1)
3. Secondary hypertension patients: Secondary hypertension is not limited to the following diseases; (e.g., renovascular disease, adrenal medullary and cortical hyperfunctions, coarctation of the aorta, hyperaldosteronism, unilateral or bilateral renal artery stenosis, Cushing's syndrome, pheochromocytoma, and polycystic kidney disease)
4. Uncontrolled diabetes mellitus (currently on insulin, or HbA1c >9% at the pre-baseline visit (V2)), or uncontrolled hypothyroidism (TSH ≥1.5 times the upper limit of normal at the pre-baseline visit (V2))
5. Heart disease (heart failure of New York Heart Association (NYHA) class 3 and 4), or ischemic heart disease (angina pectoris, myocardial infarction), peripheral vascular disease, percutaneous transluminal coronary angioplasty, or coronary artery bypass graft, etc. within 6 months prior to the screening visit (V1)
6. Clinically significant ventricular tachycardia, atrial fibrillation, atrial flutter; or other arrhythmia conditions that are determined to be clinically significant by the investigator
7. Hypertrophic obstructive cardiomyopathy, severe obstructive coronary artery disease, aortic stenosis, or hemodynamically significant aortic valve stenosis or mitral valve stenosis
8. Cerebrovascular disorder (stroke, cerebral infarction, transient cerebral ischemic attack, cerebral hemorrhage, etc. within 6 months prior to the screening visit (V1)
9. Pregnant or lactating women
10. Planning pregnancy during the study period or have childbearing potential but are not using acceptable contraceptive methods (Contraceptive methods: Refer to Section 10.1 in this document.)

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2017-05-29 (Actual); Primary Completion 2018-12-07 (Actual); Study Completion 2018-12-07 (Actual)

PRIMARY OUTCOMES:
LDL-C | 8weeks from Baseline Visit
  The percent change in LDL-C from baseline in the test group at Week 8 compared to the fimasartan 60 mg/amlodipine 10 mg combination treatment group
Sitting systolic blood pressure(SiSBP) | 8weeks from Baseline Visit
  The change in Sitting systolic blood pressure(SiSBP) from baseline in the test group at Week 8 compared to the fimasartan 60 mg and rosuvastatin 20 mg concomitant treatment group

SECONDARY OUTCOMES:
Sitting systolic blood pressure(SiSBP) | 8weeks from Baseline Visit
  The change in Sitting systolic blood pressure(SiSBP) from baseline in the test group at Week 8 compared to the fimasartan 60 mg/amlodipine 10 mg combination treatment group
LDL-C | 8weeks from Baseline Visit
  The percent change in LDL-C from baseline in the test group at Week 8 compared to the fimasartan 60 mg and rosuvastatin 20 mg concomitant treatment group

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Jeon ES, Lim SW, Kim SY, Yang HM, Kim MH, Rhee MY, Han SH, Shin J, Kim KI, Jeong JO, Sung KC, Hong GR, Kim HS, Kwon K, Kang TS, Lee HY, Han SE. A randomized, double-blind, multicenter, phase III study on the efficacy and safety of a combination treatment involving fimasartan, amlodipine, rosuvastatin in patients with essential hypertension and dyslipidemia who fail to respond adequately to fimasartan monotherapy. Clin Hypertens. 2022 Dec 1;28(1):40. doi: 10.1186/s40885-022-00223-4. PMID 36451242